CLINICAL TRIAL: NCT06871761
Title: A Randomized, Open-label, Parallel, Treat to Target Study Comparing the Efficacy and Safety of HR17031 Injection With Insulin Glargine in Patients With Type 2 Diabetes Inadequately Controlled With Basal Insulin, Metformin in Combination With or Without One Other Oral Antidiabetic Drug (OAD)
Brief Title: A Trial Comparing HR17031 With Insulin Glargine in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR17031-302
Record Dates: First submitted 2025-02-26; First posted 2025-03-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-02

CONDITIONS: Adult Patients With Type 2 Diabetes
MeSH Terms: interventions — Insulin Glargine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A: HR17031 injection (Experimental)
  Interventions: Drug: HR17031 injection
- Treatment group B: insulin glargine (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: HR17031 injection — HR17031 injection
  Arms: Treatment group A: HR17031 injection
Drug: insulin glargine — insulin glargine
  Arms: Treatment group B: insulin glargine

SUMMARY:
To compare the efficacy and safety of HR17031 injection and insulin glargine, including the changes of efficacy indicators such as HbA1c, fasting blood glucose, body weight and safety indicators such as adverse events and hypoglycemic events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18-75 years at the time of signing the informed consent (both ends included)
2. Body Mass index (BMI) of 20.0-40.0 kg/m2 (both ends included)
3. Diagnosed with type 2 diabetes for at least 90 days prior to screening
4. Tested by local laboratory, HbA1c is 7.5%-10.5% (including both ends)
5. Before screening, the daily basal insulin dose had been stabilized at 20-40U/ day (including both ends) for at least 60 days
6. Stable treatment with metformin alone or in combination with another OAD for ≥60 days prior to screening. Metformin dose ≥1500 mg/ day or maximum tolerated dose.
7. Ability and willingness to comply with protocol requirements, including self-monitoring of blood glucose, recording subject diary, and using pre-filled injection pen.

Exclusion Criteria:

1. Known or suspected allergy to the investigational drug product or its components or excipients;
2. Systemic glucocorticoid use within 3 months prior to screening
3. Use of weight loss drugs within 3 months prior to screening
4. Insulin therapy other than basal insulin was used within 3 months prior to screening
5. Cardiovascular disease, defined as congestive heart failure (NYHA III-IV), unstable angina pectoris, stroke (except lacunar infarction without symptoms), myocardial infarction, coronary revascularization within 6 months prior to screening; And/or coronary, carotid, or peripheral arterial revascularization is planned at screening
6. (with or without treatment) uncontrolled severe hypertension (systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥100 mmHg)
7. Proliferative retinopathy or macular degeneration requiring acute treatment, painful diabetic neuropathy, diabetic foot ulcers, intermittent claudication at screening;
8. Patients diagnosed with mental disorders; Mentally incapacitated or speech impediment, unable to fully understand the trial protocol or unwilling to collaborate;
9. Known or suspected abuse of alcohol or narcotics;
10. Previous history of pancreatitis (acute or chronic)
11. During pregnancy or lactation;fertile women (WOCBP) or men who have fertility plan or unwilling to use appropriate contraceptive methods from the signing of the informed consent to 3 months after last use of the investigational drug product;
12. Any condition, determined by the investigator, interfere with the efficacy or safety results of the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Changes in HbA1c from baseline to week 26 | from baseline to week 26

SECONDARY OUTCOMES:
Proportion of subjects achieved HbA1c<7.0% at week 26 | at week 26
Change in body weight from baseline to week 26 | from baseline to week 26
Proportion of subjects achieved HbA1c<7.0% and no weight gain at week 26 | at week 26
Daily Insulin dose at week 26 | at week 26
The proportion of subjects achieved HbA1c≤6.5% at week 26 | at week 26
Changes in FPG from baseline to week 26 | from baseline to week 26
Hypoglycemic event from screening to week 27 | from screening to week 27
Adverse events from screening to week 27 | from screening to week 27

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhu Xianyi Memorial Hospital, Tianjin Medical University, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided